CLINICAL TRIAL: NCT02642653
Title: Combining Lovastatin and a Parent-Implemented Language Intervention in a Multimodal Treatment for Fragile X Syndrome
Brief Title: Combining Lovastatin and a Parent-Implemented Language Intervention for Fragile X Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 520144
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Fragile X Syndrome; Genetic Diseases
Keywords: Fra(X) Syndrome; Trinucleotide Repeat Expansion; Fragile X Syndrome; Fragile X Mental Retardation Syndrome; Intellectual Disability; Parent Implemented Language Intervention (PILI); FXS; Mental Retardation, X-linked; Genetic Diseases, X-linked; Neurobehavioral Manifestations; Chromosome Disorders
MeSH Terms: conditions — Fragile X Syndrome; Genetic Diseases, Inborn; Intellectual Disability; X-Linked Intellectual Disability; Genetic Diseases, X-Linked; Neurobehavioral Manifestations; Chromosome Disorders | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lovastatin and PILI (Active Comparator): Subjects will receive the Parent Implemented Language Intervention (PILI) in combination with study medication Lovastatin.
  Interventions: Drug: Lovastatin
- Placebo and PILI (Placebo Comparator): Subjects will receive the Parent Implemented Language Intervention (PILI) in combination with placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lovastatin — Once per day dosing
  Other Names: Mevacor
  Arms: Lovastatin and PILI
Other: Placebo — Once per day dosing
  Arms: Placebo and PILI

SUMMARY:
The purpose of the study is to test the efficacy of a 20 week multi-modal treatment comprised of lovastatin or placebo, and the Parent-implemented Language Intervention (PILI) in children with fragile X syndrome (FXS). Children will be randomized to drug or placebo in a double-blind design with all participating in the PILI. The primary endpoint will be to measure improvements in spoken language and behavior among lovastatin-treated than placebo treated participants.

DETAILED DESCRIPTION:
This is the first multi-modal treatment to combine a targeted treatment for FXS, lovastatin, with an innovative parent-implemented intervention (PILI) targeting language and challenging behavior delivered through telehealth technology.The hypothesis is that targeted treatments will be more effective when applied in combination with PILI. Examination of whether changes in the activity of key pathways/proteins influenced by fragile X mental retardation protein (FMRP) (the mitogen-activated protein kinase (ERK) and MMP-9) are biomarkers of treatment responsiveness. Because lovastatin is also an anti-inflammatory, characterization of MEK/ERK signaling in peripheral immune cells both pre- and post- treatment will be carried out to determine whether levels of these signaling molecules are predictive biomarkers of treatment response. It is hypothesized that those individuals with elevated inflammatory cytokine profiles will be most responsive to lovastatin treatment. Once modeled in FXS, results from these studies can then be applied to other neurodevelopmental disorders including RASopathies.

The behavioral component of the proposed multi-modal treatment will be a Parent-implemented Intervention (PILI) that targets improvements in spoken language and challenging behavior for 10- to 17-year-olds with FXS by increasing parental verbal responsiveness (PVR) within picture-book based story-telling episodes. Parents will be encouraged to use the targeted strategies in other everyday interactions with their child. The intervention will be delivered to parents in their homes by way of video teleconferencing (VTC). Participants will be randomly assigned to receive the behavioral intervention alone or in combination with Lovastatin.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a full mutation with absence or deficient FMRP levels.
* Males and females ages 10 through 17 years
* Willingness of potential study participant as well as a parent or caretaker to participate in the protocol.
* Speech is the primary means of communication with three-word or longer utterances used on a daily basis.
* Intelligence quotient (IQ) ≤70 as measured by the Leiter- R.
* Sexually active women of childbearing potential (WCBP) must be using a medically acceptable method of birth control and have a negative qualitative serum β-human chorionic growth hormone (β-HCG) or urine pregnancy test collected at the initial screening visit.

Exclusion Criteria:

* Persons who do not speak English.
* Changes in any medications (including investigational medications) within the last month (4 weeks). All concomitant medications must have been on a stable course for at least 4 weeks prior to enrollment into the study and maintain stability throughout the course of the study.
* Changes in behavioral therapy or educational programming during the study. This does not include scheduled school holidays.
* Have any disease or condition (medical or surgical) at screening that might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or hepatic systems; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the investigational product, or would place the subject at increased risk.
* Patients who, in the opinion of the investigator, are unsuitable in any other way to participate in this study, including being unable to comply with the requirements of the study or displaying clinically significant abnormalities in safety assessments at screening.
* Patients on prohibited medications
* History of recurrent status epilepticus.
* Inability to withhold grapefruit and grapefruit juice from diet during the entire clinical trial.
* Subjects unwilling to abstain from alcoholic beverages during the trial.
* Subjects who are actively suicidal.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurman AJ, Potter LA, Kim K, Tassone F, Banasik A, Potter SN, Bullard L, Nguyen V, McDuffie A, Hagerman R, Abbeduto L. Controlled trial of lovastatin combined with an open-label treatment of a parent-implemented language intervention in youth with fragile X syndrome. J Neurodev Disord. 2020 Apr 22;12(1):12. doi: 10.1186/s11689-020-09315-4. PMID 32316911

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lovastatin and PILI | Placebo and PILI
Started | 14 | 16
Completed | 12 | 16
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lovastatin and PILI | Placebo and PILI | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 16 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.86 (2.14) | 13.17 (2.54) | 13.52 (2.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 10 | 24
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Intelligence Quotient (IQ) [Mean (Standard Deviation); unit: units on a scale] — A standardized test designed to measure developmental functioning and IQ for individuals ranging in age from 2 years to adulthood. Minimal verbal directions are used in the administration to allow assessment of cognitive ability independent of language ability. The Brief IQ screener is composed of 4 subtests: figure ground, form completion, sequential order, and repeated patterns subtests. IQ scores are the sum of the scaled scores for the subtests. Scores range from a minimum of 36 to a maximum of 169.
  units on a scale | 44.00 (9.22) | 43.13 (6.24) | 43.57 (7.73)
Cognitive growth score [Mean (Standard Deviation); unit: units on a scale] — Growth Scores are useful for the interpretation of an individual child's performance. Since the child's overall ability level is placed along a linear scale. Raw scores for each Leiter-R subtest are converted into Growth Scale Scores. The score is a three-digit number that can range from 380 to 560. Higher scores represent higher ability levels.
  units on a scale | 461.4 (13.32) | 462.3 (8.57) | 461.85 (10.95)
Autism Diagnostic Observation Scale (ADOS) severity score [Mean (Standard Deviation); unit: units on a scale] — The Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) The assessment will provide a continuous metric of autism symptom severity for use in characterizing the participant sample and as a potential moderator of treatment response. The ADOS is a gold-standard measure of current symptoms of autism. Total scores will be used to assign a severity score. Scores range from 1 to 10, with higher scores reflecting more severe impairment
  units on a scale | 6.85 (2.54) | 6.75 (2.05) | 6.80 (2.30)

OUTCOME MEASURES:

1. Primary Outcome: Expressive Language Sample Composite Score in the Home
Description: The primary outcome reflects the diversity of vocabulary used. Higher scores reflect more skill. The lowest possible value is zero. No theoretical maximum can be defined because the wordless picture books can lead to a large and indeterminate set of options for the amount of talk and the vocabulary used. In a previous study of a nonpharmacological intervention, the range at baseline was 9-177, and at post-treatment, the range for the combined treated and nontreated groups was 23-214, although these values were not corrected for the number of C-units produced (McDuffie at el. 2018 Developmental Neurorehabilitation).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
score on a scale | 39.63 (32.41) | 42.47 (18.60)

2. Secondary Outcome: FXS- Normed Aberrant Behavior Checklist (ABC) Social Avoidance Subscale
Description: The ABC-C is a 58-item caregiver-rated behavior scale used to examine treatment effects on challenging behaviors for individuals with FXS in the following domains: (1) irritability; (2) lethargy/social withdrawal; (3) stereotypic behavior; (4) hyperactivity; and (5) inappropriate speech. Caregiver rates the subject's behavior as follows: 0 = not a problem, l = the behavior is a problem but slight in degree, 2 = the problem is moderately serious, 3 = the problem is severe in degree. Sansone et al. (2012) further subdivided social withdrawal to rate social avoidance in FXS. The subscale includes 4 items which were originally part of the Lethargy/Withdrawal subscale. This subscale captures core aspects of the FXS phenotype related to gaze avoidance, social ''escape'' behaviors, and social anxiety. Subscale score ranges from 0 to 12, higher scores reflect a more problematic behavior.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
score on a scale | 2.5 (2.84) | 4.31 (3.66)

3. Secondary Outcome: FXS- Normed Aberrant Behavior Checklist (ABC) Social Avoidance Subscale
Description: The ABC-C is a 58-item caregiver-rated behavior scale used to examine treatment effects on challenging behaviors for individuals with FXS in the following domains: (1) irritability; (2) lethargy/social withdrawal; (3) stereotypic behavior; (4) hyperactivity; and (5) inappropriate speech. Caregiver rates the subject's behavior as follows: 0 = not a problem, l = the behavior is a problem but slight in degree, 2 = the problem is moderately serious, 3 = the problem is severe in degree. Sansone et al. (2012) further subdivided social withdrawal to rate social avoidance in FXS. The subscale includes 4 items which were originally part of the Lethargy/Withdrawal subscale. This subscale captures core aspects of the FXS phenotype related to gaze avoidance, social ''escape'' behaviors, and social anxiety. Subscale score ranges from 0 to 12, higher scores reflect a more problematic behavior. Shown here are the ABC social avoidance subscale mean scores from the 10-weeks follow-up visit.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
score on a scale | 2.5 (2.11) | 3.53 (3.68)

4. Secondary Outcome: FXS- Normed Aberrant Behavior Checklist (ABC) Social Avoidance Subscale
Description: The ABC-C is a 58-item caregiver-rated behavior scale used to examine treatment effects on challenging behaviors for individuals with FXS in the following domains: (1) irritability; (2) lethargy/social withdrawal; (3) stereotypic behavior; (4) hyperactivity; and (5) inappropriate speech. Caregiver rates the subject's behavior as follows: 0 = not a problem, l = the behavior is a problem but slight in degree, 2 = the problem is moderately serious, 3 = the problem is severe in degree. Sansone et al. (2012) further subdivided social withdrawal to rate social avoidance in FXS. The subscale includes 4 items which were originally part of the Lethargy/Withdrawal subscale. This subscale captures core aspects of the FXS phenotype related to gaze avoidance, social ''escape'' behaviors, and social anxiety. Subscale score ranges from 0 to 12, higher scores reflect a more problematic behavior. Shown are the ABC social avoidance subscale mean scores from the 20-weeks end-of-study visit.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
score on a scale | 2.42 (2.84) | 3.38 (3.34)

5. Secondary Outcome: Clinical Global Impression- Severity (CGI-S)
Description: A clinician rated scale utilizing history from the parents or caregiver and incorporating it into a clinical rating for severity. The CGI-S was used at the pre-treatment assessment to judge symptom severity. The 7-point scale ranges from: 1 = Normal; 2 = Borderline Ill; 3 = Mildly Ill; 4 = Moderately Ill; 5 = Markedly Ill; 6 = Severely Ill; and 7 = Extremely Ill. Therefore, the higher the score, the greater the severity of the patient's illness. Shown here are the CGI-S mean scores from the baseline visit.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
units on a scale | 4.58 (0.67) | 4.50 (0.63)

6. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Scale
Description: A clinician rated scale utilizing history from the parents or caregiver and incorporating it into a clinical rating to assess for overall therapeutic response. The 7-point scale ranges from: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse. Therefore, the lower the score, the greater the overall improvement as rated by the clinician. The CGI-I was used at the 10 week and 20 week visits. Shown here are the CGI-I mean scores from the 10-weeks end-of-study visit.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
units on a scale | 2.92 (0.79) | 3.00 (0.73)

7. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Scale
Description: A clinician rated scale utilizing history from the parents or caregiver and incorporating it into a clinical rating to assess for overall therapeutic response. The 7-point scale ranges from: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse. Therefore, the lower the score, the greater the overall improvement as rated by the clinician. The CGI-I was used at the 10 week and 20 week visits. Shown here are the CGI-I mean scores from the 20-weeks end-of-study visit.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
units on a scale | 2.42 (0.67) | 2.38 (0.72)

8. Secondary Outcome: Visual Analog Scale (VAS) - Spoken Language Impairment
Description: The measure was used to assess parental impressions of progress in two key symptoms: spoken language impairment and social impairment. The distance of the mark from one end is used as the outcome variable for analysis. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 10-weeks and 20-weeks visits. The calculated distance in cm between the marks drawn at the baseline and follow-up visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Spoken Language Impairment scale, at baseline. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
centimeters | 4.06 (2.43) | 1.94 (1.41)

9. Secondary Outcome: Visual Analog Scale (VAS) - Spoken Language Impairment
Description: The measure was used to assess parental impressions of progress in two key symptoms: spoken language impairment and social impairment. The distance of the mark from one end is used as the outcome variable for analysis. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 10-weeks and 20-weeks visits. The calculated distance in cm between the marks drawn at the baseline and follow-up visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Spoken Language Impairment scale, at 10-weeks. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
centimeters | 5.28 (2.69) | 3.09 (1.14)

10. Secondary Outcome: Visual Analog Scale (VAS) - Spoken Language Impairment
Description: The measure was used to assess parental impressions of progress in two key symptoms: spoken language impairment and social impairment. The distance of the mark from one end is used as the outcome variable for analysis. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 10-weeks and 20-weeks visits. The calculated distance in cm between the marks drawn at the baseline and follow-up visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Spoken Language Impairment scale, at 20-weeks. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
centimeters | 5.66 (1.99) | 4.18 (1.53)

11. Secondary Outcome: Visual Analog Scale (VAS) - Social Impairment
Description: The measure was used to assess parental impressions of progress in two key symptoms: spoken language impairment and social impairment. The distance of the mark from one end is used as the outcome variable for analysis. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 10-weeks and 20-weeks visits. The calculated distance in cm between the marks drawn at the baseline and follow-up visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Social Impairment scale, at baseline. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
centimeters | 3.73 (1.74) | 2.55 (1.36)

12. Secondary Outcome: Visual Analog Scale (VAS) - Social Impairment
Description: The measure was used to assess parental impressions of progress in two key symptoms: spoken language impairment and social impairment. The distance of the mark from one end is used as the outcome variable for analysis. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 10-weeks and 20-weeks visits. The calculated distance in cm between the marks drawn at the baseline and follow-up visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Social Impairment scale, at 10-weeks. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: 10-weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
centimeters | 4.57 (2.15) | 3.41 (1.61)

13. Secondary Outcome: Visual Analog Scale (VAS) - Social Impairment
Description: The measure was used to assess parental impressions of progress in two key symptoms: spoken language impairment and social impairment. The distance of the mark from one end is used as the outcome variable for analysis. Caregivers mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 10-weeks and 20-weeks visits. The calculated distance in cm between the marks drawn at the baseline and follow-up visits thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side for the Social Impairment scale, at 20-weeks. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
centimeters | 5.18 (1.70) | 3.99 (2.06)

14. Primary Outcome: Expressive Language Sample Composite Score in the Home
Description: as for outcome 1
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lovastatin and PILI | Placebo and PILI
Number analyzed (Participants) | 12 | 16
score on a scale | 59.32 (22.81) | 54.81 (16.04)

ADVERSE EVENTS:
Time Frame: From baseline to follow-up (20-weeks)
Arm/Group | Lovastatin and PILI | Placebo and PILI
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 11/12 | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin and PILI (N=12) | Placebo and PILI (N=16)
Abnormal vocalizations (Psychiatric disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Decreased Appetite (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Disruptive behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry Mouth (Nervous system disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Elevated Bilirubin (Hepatobiliary disorders) | 0 (0) | 1 (1)
Emotional Lability (Psychiatric disorders) | 0 (0) | 2 (2)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Eye Infection (Eye disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (2) | 0 (0)
Gastrointestinal issues (Gastrointestinal disorders) | 2 (2) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hyperactivity (Psychiatric disorders) | 2 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Menstrual Cramps (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Obsessive compulsive behavior (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Self-injurious behavior (Psychiatric disorders) | 0 (0) | 1 (1)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Skin_Infection (Infections and infestations) | 1 (2) | 2 (2)
Sleep Disturbance (Psychiatric disorders) | 1 (1) | 1 (1)
Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 7 (10) | 8 (12)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study did not have a cohort treated only with lovastatin without the parent-implemented language intervention (PILI). The efficacy of the study medication alone compared to placebo can't be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT02642653/Prot_SAP_000.pdf